CLINICAL TRIAL: NCT02289755
Title: A Phase 2 Multicenter, Open Label, Single Arm Study Evaluating the Effect of ALLN-177 to Reduce Urinary Oxalate Excretion in Recurrent Calcium Oxalate Kidney Stone Formers With Hyperoxaluria
Brief Title: Evaluating ALLN-177 for Reducing Urinary Oxalate Excretion in Calcium Oxalate Kidney Stone Formers With Hyperoxaluria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0000396
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2016-02

CONDITIONS: Hyperoxaluria; Nephrolithiasis
Keywords: Urine Oxalate; Nephrolithiasis; Kidney Stones; Hyperoxaluria; Enteric Hyperoxaluria; Idiopathic Hyperoxaluria; Urological Diseases; Kidney Diseases
MeSH Terms: conditions — Hyperoxaluria; Nephrolithiasis; Kidney Calculi; Urologic Diseases; Kidney Diseases | interventions — reloxaliase; oxalate decarboxylase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALLN-177 (Experimental): Recurrent Calcium Oxalate Stone Formers with Hyperoxaluria Subjects with Enteric or Idiopathic hyperoxaluria
  Dosing: 5 capsules of ALLN-177 orally (p.o.) up to 3 times daily (TID) with meals for 4 consecutive days.
  Interventions: Drug: ALLN-177

INTERVENTIONS:
Drug: ALLN-177 — ALLN-177 is orally administered oxalate decarboxylase (OxDc). The goal of oral therapy with ALLN-177 is to enzymatically degrade both dietary oxalate and endogenously produced oxalate secreted in the gastrointestinal tract resulting in decreased absorption and reduced urinary oxalate excretion.
  Other Names: Oxalate degrading enzyme; Oxalate decarboxylase

SUMMARY:
The purpose of this study is to evaluate the effect of ALLN-177 to reduce urinary oxalate excretion in patients with recurring kidney stones and enteric or idiopathic hyperoxaluria.

DETAILED DESCRIPTION:
A multi-center, open-label, single arm study to evaluate the safety and the effect of ALLN-177 to reduce urinary oxalate excretion in recurrent kidney stone formers with associated hyperoxaluria. The study design includes a screening period to confirm eligibility, followed by a 3-day baseline period, 4-day open label treatment period with ALLN-177 and 4-day follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Able to comply with study procedures
* History of enteric or idiopathic hyperoxaluria and at least one calcium oxalate kidney stone
* Hyperoxaluria >36mg of oxalate/24-hr
* May be taking drugs for the prevention of stone disease as long as there have been no changes in these medications for at least 3 months

Exclusion Criteria:

* Uric acid ≥1.5g/24-hr
* Estimated glomerular filtration rate of < 60 mL/min
* Positive results from drug urine screen
* Requires daily vitamin C (defined as >10 days of >300 mg/day)
* Diagnosis of hypercalcemia or hypothyroidism
* Obstructive uropathy, chronic urosepsis, renal failure, renal tubular acidosis, primary hyperparathyroidism, primary hyperoxaluria, pure uric acid and cystine stones, and/or medullary sponge kidney.
* Auto-immune disorder requiring high dose steroids or other immunosuppressant drugs.
* Subjects who are pregnant. Women of childbearing potential must have a negative pregnancy test prior to enrollment and must practice approved methods of birth control during the trial
* History of cancer diagnosis except for within the past 5 years excluding dermal squamous and/or basal cell carcinoma or cervical carcinoma in situ.
* Taken investigational compound within 30 days prior to the first day of the study
* Treatment with cholestyramine
* Average daily dietary intake of <75 mg oxalate per day calculated from diet recalls

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Brettman, MD, FACP, Study Director — Medical Director
Locations (4):
- United States (4):
  - Indiana University Physicians Urology, Indianapolis, Indiana
  - North Shore Long Island Jewish Health System, Lake Success, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Omega Clinical Research, Warwick, Rhode Island

REFERENCES:
- [Derived] Lingeman JE, Pareek G, Easter L, Pease R, Grujic D, Brettman L, Langman CB. ALLN-177, oral enzyme therapy for hyperoxaluria. Int Urol Nephrol. 2019 Apr;51(4):601-608. doi: 10.1007/s11255-019-02098-1. Epub 2019 Feb 19. PMID 30783888

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects (N = 16) were recruited from 3 centers in the United States between August 2014 and December 2014.
Pre-assignment Details: History of ≥1 calcium oxalate kidney stone within the last 2 years, secondary hyperoxaluria and a mean urinary oxalate of ≥36 mg/day
Groups:
- ALLN-177: ALLN-177 (5 capsules; 7,500 units/meal) by mouth 3 times a day with main meals for 4 consecutive days.
Period: Baseline Period [No Treatment, 3 Days]
Arm/Group | ALLN-177
Started | 16
Completed | 16
Not Completed | 0
Period: ALLN-177 Treatment Period [4 Days]
Arm/Group | ALLN-177
Started | 16
Completed | 16
Not Completed | 0
Period: Follow up Period [4 Days]
Arm/Group | ALLN-177
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects (N=16) were included in the analysis.
Groups:
- ALLN-177: ALLN-177 (5 capsules: 7,500 units/meal), 3 times a day with meals, 4 days
Arm/Group | ALLN-177
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (14.5)
Age, Continuous [Median (Full Range); unit: years] | 58.0 [24 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Glomerular Filtration Rate (GFR) [Mean (Full Range); unit: ml/min/1.73 m^2] | 85.1 [39 to 118]
Concomitant medications [Number; unit: participants] — Usual methods for treatment of kidney stones/nephrolithiasis were continued throughout the study. Participants could have been prescribed more than one medication, so the sum of participants would be greater than the population.
  participants
    Potassium citrate | 5
    Chlorthalidone | 2
    Hydrochlorothiazide | 1
    Calcium | 5
24-hour Urinary Oxalate [Mean (Standard Deviation); unit: mg/day] | 77.65 (55.87)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Period to Treatment Period 24-hour Urinary Oxalate Excretion
Description: Change from Baseline is defined as Baseline value (average of Days 2 and 3) minus ALLN-177 treatment value (mean of Days 5, 6, and 7).
Time Frame: 7 days
Population: All Participants (N=16) completed treatment and were included in the analysis population.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | ALLN-177
Number analyzed (Participants) | 16
mg/day | -13.92 (18.37)

2. Secondary Outcome: Percent Change From Baseline Period to Treatment Period in 24-hour Urinary Oxalate Excretion
Description: Percent Change from Baseline is defined as baseline value (average of Days 2 and 3) minus ALLN-177 treatment value (mean of Days 5, 6, and 7) divided by baseline value times 100%
Time Frame: 7 days
Population: All Participants (N=16) were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | ALLN-177
Number analyzed (Participants) | 16
percentage change | -13.28 (16.62)

ADVERSE EVENTS:
Time Frame: Up to 11 days.
Description: Treatment-emergent adverse events = AEs with onset at or after starting study drug through 7 days after the last dose of study drug.
Arm/Group | ALLN-177
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 9/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALLN-177 (N=16)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days